CLINICAL TRIAL: NCT06732115
Title: Esthetic Performance and Surface Roughness of Class IV Nanohybrid Composite Restorations Following One-step Versus Multistep Polishing Protocol: a Randomized Clinical Trial
Brief Title: Effect of One-step Versus Multistep Polishing Protocol on Class IV Composite Restorations.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noreen Amr Labib, Master degree student in operative department, faculty of dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230084
Record Dates: First submitted 2024-12-06; First posted 2024-12-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-12

CONDITIONS: Esthetic Restorations
Keywords: Surface roughness; class IV; nanohybrid composite; multistep polishing system.; one-step polishing system; surface staining

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): One-step polishing system with nanohybrid resin composite restorations
  Interventions: Procedure: One-step polishing system with nanohybrid resin composite restorations.
- Compartor (Active Comparator): Multistep system polishing system with nanohybrid resin composite restorations.
  Interventions: Procedure: Multistep system polishing system Super-Snap X-treme (Shofu) with nanohybrid resin composite restorations.

INTERVENTIONS:
Procedure: One-step polishing system with nanohybrid resin composite restorations. — one-step polishing system using OneGloss by Shofu
  Arms: Intervention
Procedure: Multistep system polishing system Super-Snap X-treme (Shofu) with nanohybrid resin composite restorations. — A multi-step polishing system
  Arms: Compartor

SUMMARY:
This study aims to evaluate the effectiveness of various finishing and polishing techniques for composite resins used in dental restorations, with a focus on minimizing discoloration and surface roughness over time. Discoloration due to plaque accumulation and surface staining can lead to esthetic concerns, resulting in premature restoration replacement and increased costs. Prior research highlights that esthetic failures, such as color alterations and surface staining, are key reasons for the failure of anterior restorations. Given the contradictory findings in previous studies on finishing and polishing methods, this research seeks to determine whether one-step polishing system will have the same effect as the multistep system in terms of esthetic performance and surface roughness of nanohybrid resin composite class IV restorations. The main operator will compare between OneGloss (Shofu) the intervention and Super-Snap X-treme (Shofu) the comparator. Patients will be evaluated immediately following polishing then after 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient related criteria:

  * Patients with good general health.
  * Patients who agreed to the consent and committed to follow-up period
  * No specific age range.
  * Both genders.
  * Low and moderate caries risk patients
  * Normal occlusion
* Tooth related criteria

  * Fully erupted permanent anterior teeth with class IV.
  * Active caries, fractures, or defective Restorations in anterior teeth.

Exclusion Criteria:

* Patient related criteria

  * Patient with bad oral hygiene.
  * Patients with tetracycline or fluorosis staining.
  * Patients who could/would not participate in all times of follow-up.
  * Patients participating in more than 1 dental study.
  * Patient received fluoride varnish, or during orthodontic treatment.
  * Patients with tendency to do bleaching during the study.
  * Heavy Smokers
  * Patients who are alcoholic and addicted Tooth related criteria
  * Untreated periodontal disease was not allowed
  * Fully erupted anterior teeth with no defects

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Surface Luster (success rate) | 24hours, 3 months, 6months and 12 months
  Scoring system (ordinal) 5: Luster comparable to enamel 4: Slightly dull, not noticeable from speaking distance, some isolated pores 3: Dull surface but acceptable if covered with film of saliva, multiple pores on more that one-third of the surface 2: Rough surface, cannot be masked by saliva film, simple polishing not sufficient
  1: Very rough, unacceptable plaque-retentive surface

SECONDARY OUTCOMES:
Surface Staining | 24hours, 3 months, 6months and 12 months
  Scoring system (ordinal) 5: No staining 4: Minor Staining, easily removable by polishing 3: Moderate surface staining that may also be present on other teeth, not esthetically unacceptable 2: Unacceptable surface staining, major intervention necessary
  1: severe surface and/or subsurface staining, not acceptable for intervention
Marginal Staining | 24hours, 3 months, 6months and 12 months
  Scoring system (ordinal) 5 No staining 4 Minor staining, easily removable by polishing 3 Moderate marginal staining, not esthetically unacceptable 2 Pronounced marginal staining; major intervention necessary
  1 Deep marginal staining, not accessible for intervention
Color Match | 24hours, 3 months, 6months and 12 months
  Scoring system (ordinal)
  1. Good color match, no difference in shade and translucency
  2. Minor Deviation
  3. Clear deviation but acceptable. Does not affect esthetic 3.1: More opaque 3.2: More translucent 3.3: Darker 3.4: Brighter
Surface Roughness | 24hours, 3 months, 6months and 12 months
  Surface roughness means (Ra)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No